CLINICAL TRIAL: NCT00556322
Title: An Open-label, Randomized Study to Evaluate the Effect of Tarceva, Compared With Alimta (Pemetrexed) or Taxotere (Docetaxel),on Survival in Patients With Advanced, Recurrent or Metastatic Non-small Cell Lung Cancer Who Have Experienced Disease Progression During Platinum-based Chemotherapy
Brief Title: A Study of Tarceva (Erlotinib) and Standard of Care Chemotherapy in Patients With Advanced, Recurrent, or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO18602
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Docetaxel; Erlotinib Hydrochloride

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]
- 2 (Active Comparator)
  Interventions: Drug: Alimta or Taxotere

INTERVENTIONS:
Drug: Alimta or Taxotere — 500mg/m2 / 3 weeks (Alimta) or 75mg/m2 / 3 weeks (Taxotere)
  Arms: 2
Drug: erlotinib [Tarceva] — 150mg po daily
  Arms: 1

SUMMARY:
This 2 arm study will evaluate the efficacy, safety, and pharmacokinetics of Tarceva and that of standard of care chemotherapy in patients with advanced, recurrent, or metastatic NSCLC experiencing disease progression after failure of platinum-based chemotherapy.Eligible patients will be randomized to receive either Tarceva 150mg po daily, or comparator (either Alimta 500mg/m2 every 3 weeks, or Taxotere 75mg/m2 every 3 weeks). The anticipated time on study treatment is until disease progression ,and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* histologically documented, locally advanced or recurrent or metastatic NSCLC;
* measurable disease;
* disease progression during 1-4 cycles of platinum-based chemotherapy.

Exclusion Criteria:

* any other malignancies within the last 5 years;
* unstable systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2006-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (106):
- Australia (7):
  - St Leonards, New South Wales
  - Waratah, New South Wales
  - Adelaide, South Australia
  - East Bentleigh, Victoria
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
- Austria (3):
  - Innsbruck
  - Klagenfurt
  - Vienna
- Antwerp, Belgium
- Canada (6):
  - Winnipeg, Manitoba
  - Oshawa, Ontario
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Montreal, Quebec
- Santiago, Chile
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai
- Czechia (3):
  - České Budějovice
  - Olomouc
  - Pilsen
- Denmark (2):
  - Herlev
  - Odense
- France (11):
  - Bayonne
  - Brest
  - Clermont-Ferrand
  - Dijon
  - Le Mans
  - Lille
  - Limoges
  - Paris
  - Pau
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Bad Berka
  - Bochum
  - Halle
  - Herne
  - Neuruppin
  - Villingen-Schwenningen
- Greece (2):
  - Athens
  - Heraklion
- Hungary (6):
  - Budapest
  - Deszk
  - Nyíregyháza
  - Pécs
  - Szombathely
  - Törökbálint
- Italy (3):
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Ancona, The Marches
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Malaysia (2):
  - George Town
  - Kuala Lumpur
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (2):
  - Lodz
  - Otwock
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Timișoara
- Russia (14):
  - Arkhangelsk
  - Balashikha
  - Chelyabinsk
  - Kazan'
  - Kirov
  - Krasnodar
  - Kuzmolovo
  - Moscow
  - Nizhny Novgorod
  - Perm
  - Saint Petersburg
  - Sashi
  - Smolensk
  - Yaroslavl
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Nitra
  - Poprad
- Slovenia (3):
  - Golnik
  - Ljubljana
  - Maribor
- South Africa (3):
  - Durban
  - Johannesburg
  - Pretoria
- South Korea (3):
  - Daegu
  - Seoul
  - Suwon
- Spain (4):
  - Santander, Cantabria
  - A Coruña, La Coruña
  - Oviedo, Principality of Asturias
  - Zaragoza, Zaragoza
- Ukraine (3):
  - Kharkiv
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (4):
  - Chelmsford
  - Dundee
  - Leicester
  - Plymouth
- Caracas, Venezuela

REFERENCES:
- [Derived] Ciuleanu T, Stelmakh L, Cicenas S, Miliauskas S, Grigorescu AC, Hillenbach C, Johannsdottir HK, Klughammer B, Gonzalez EE. Efficacy and safety of erlotinib versus chemotherapy in second-line treatment of patients with advanced, non-small-cell lung cancer with poor prognosis (TITAN): a randomised multicentre, open-label, phase 3 study. Lancet Oncol. 2012 Mar;13(3):300-8. doi: 10.1016/S1470-2045(11)70385-0. Epub 2012 Jan 24. PMID 22277837

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator: Participants received either pemetrexed 500 milligrams per square meter (mg/m^2) every 21 days until disease progression, unacceptable toxicity or death or docetaxel 75 mg/m^2 every 3 weeks until disease progression, unacceptable toxicity or death. Choice of comparator was left to the discretion of the investigator in countries where both treatments are registered to use and are commercially available for second line use (otherwise, docetaxel was administered), assigning the participant to either comparator depending upon the medical needs of the participant. Participants were required to receive concomitant treatment therapy as indicated in the product label.
- Erlotinib: Participants received erlotinib, 150 mg, administered orally as a tablet, once daily until disease progression, unacceptable toxicity, or death.
Period: Overall Study
Arm/Group | Comparator | Erlotinib
Started | 221 | 203
Completed | 0 (Data cutoff was 01 August 2010) | 0 (Data cutoff was 01 August 2010)
Not Completed | 221 | 203
Not completed — Insufficient therapeutic response | 158 | 168
Not completed — Adverse Event | 7 | 4
Not completed — Other | 4 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 19 | 7
Not completed — Protocol Violation | 5 | 1
Not completed — Ongoing at data cutoff | 3 | 5
Not completed — Death | 20 | 14

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants randomized were included according to the therapy that they were randomized to receive in the FAS population.
Groups:
- Comparator: Participants received either pemetrexed 500 mg/m^2 every 21 days until disease progression, unacceptable toxicity or death or docetaxel 75 mg/m^2 every 3 weeks until disease progression, unacceptable toxicity or death. Choice of comparator was left to the discretion of the investigator in countries where both treatments are registered to use and are commercially available for second line use (otherwise, docetaxel was administered), assigning the participant to either comparator depending upon the medical needs of the participant. Participants were required to receive concomitant treatment therapy as indicated in the product label.
- Total: Total of all reporting groups
Arm/Group | Comparator | Erlotinib | Total
Number analyzed (Participants) | 221 | 203 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.90) | 58.6 (9.64) | 58.4 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 42 | 103
  Male | 160 | 161 | 321

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died (All Participants; Data Cutoff: 07 September 2010)
Description: Overall survival (OS) was determined from the date of randomization to the date of death irrespective of the cause of death.
Time Frame: Baseline, Weeks 3 and 6, Every 3 Weeks until Week 48 or Death and Every 12 Weeks until Death or Data Cut off (07 September 2010) up to 52 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants | 81.0 | 77.8

2. Primary Outcome: Duration of Overall Survival in All Participants (Data Cutoff 07 September 2010)
Description: OS was determined from the date of randomization to the date of death irrespective of the cause of death. Kaplan-Meier estimates were used for analysis.
Time Frame: Baseline, Weeks 3 and 6, Every 3 Weeks until Week 48 and Every 12 Weeks until Death or Until Data Cut off (07 September 2010) up to 52 months
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
months | 5.5 [4.4 to 7.1] | 5.3 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.7299, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.78 to 1.19]

3. Primary Outcome: Probable Percentage of Participants Remaining Alive at 1 Year
Description: as for outcome 2
Time Frame: 1 Year
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants | 24.0 [18.0 to 30.0] | 26.0 [19.0 to 32.0]

4. Secondary Outcome: Percentage of Participants Who Died in Epidermal Growth Factor Receptor (EGFR) Positive and Negative Population
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR was determined by immunohistochemistry (IHC). OS was determined from the date of randomization to the date of death irrespective of the cause of death in EGFR positive and negative populations. Kaplan-Meier estimates were used for analysis.
Time Frame: as for outcome 2
Population: FAS population; Only participants with confirmed presence or absence of EGFR were included in the analysis. number (n) equals (=) number of participants who were EGFR positive or negative
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 188 | 175
percentage of participants
  EGFR Positive (n=149,143) | 79.9 | 76.9
  EGFR Negative (n=39,32) | 79.5 | 75.0

5. Secondary Outcome: Duration of OS in EGFR Positive and Negative Population
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR was determined by IHC. OS was determined from the date of randomization to the date of death irrespective of the cause of death in EGFR positive and negative populations. Kaplan-Meier estimates were used for analysis.
Time Frame: as for outcome 2
Population: FAS population; Only participants with confirmed presence or absence of EGFR were included in the analysis. n=number of participants who were EGFR positive or negative
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 188 | 175
months
  EGFR Positive (n=149,143) | 5.5 [4.1 to 7.5] | 5.6 [4.0 to 7.6]
  EGFR Negative (n=39,32) | 6.7 [3.1 to 11.5] | 5.4 [3.7 to 7.8]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Comparison of EGFR positive populations; Test type: Superiority or Other; p = 0.6198, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.72 to 1.21]
Statistical Analysis 2: Comparison: Comparator vs Erlotinib; Comparison of EGFR negative populations; Test type: Superiority or Other; p = 0.8398, Log Rank; Hazard Ratio, log = 0.95, 95% CI 2-sided [0.55 to 1.62]

6. Secondary Outcome: Probable Percentage of Participants Remaining Alive at 1 Year in the EGFR Positive and Negative Population
Description: as for outcome 5
Time Frame: 1 Year
Population: FAS population; n=number of EGFR positive or negative participants remaining at risk
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Comparator: Participants received either pemetrexed 500 mg/m^2 every 21 days until disease progression, unacceptable toxicity or death or docetaxel l75 mg/m^2 every 3 weeks until disease progression, unacceptable toxicity or death. Choice of comparator was left to the discretion of the investigator in countries where both treatments are registered to use and are commercially available for second line use (otherwise, docetaxel was administered), assigning the participant to either comparator depending upon the medical needs of the participant. Participants were required to receive concomitant treatment therapy as indicated in the product label.
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants
  EGFR Positive (n=30,32) | 27.0 [19.0 to 34.0] | 30.0 [22.0 to 38.0]
  EGFR Negative (n=8,4) | 28.0 [12.0 to 43.0] | 20.0 [4.0 to 36.0]

7. Secondary Outcome: Percentage of Participants With Disease Progression or Death (All Participants; Data Cut Off 07 September 2010)
Description: Tumor response was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.0). Progressive Disease was defined as at least a 20 percent (%) increase in the sum of the Longest Diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The primary analysis of PFS used objective progression (RECIST) plus clinical progression (based on relevant clinical findings - if any). A further assessment of PFS was made on objective (radiological) progression. If clinical progression was diagnosed first, the participant was censored at the date of the last tumor assessment, where non-progression was documented.
Time Frame: Baseline, Weeks 3 and 6, Every 3 Weeks until Week 48 and Every 12 Weeks until Disease Progression or unacceptable toxicity or Until Data Cut off (07 September 2010) up to 52 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants | 83.3 | 92.6

8. Secondary Outcome: Progression-Free Survival (PFS) in All Participants (Data Cutoff 07 September 2010)
Description: Tumor response was evaluated according to RECIST criteria (version 1.0). Progressive Disease was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PFS was defined as time from randomization to the date of documented disease progression or death, whichever occurred first. Participants without progression were censored at the date of last tumor assessment where non progression was documented. If a participant receives a second anti-cancer therapy without prior documentation of disease progression, the participant was censored at the date of last tumor assessment before starting new chemotherapy.
Time Frame: as for outcome 7
Population: FAS population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
weeks | 8.6 [7.1 to 12.1] | 6.3 [6.1 to 6.9]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.0885, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.97 to 1.46]

9. Secondary Outcome: Probable Percentage of Participants Remaining Alive and Progression Free at 6 Months
Description: Tumor response was evaluated according to RECIST criteria (version 1.0). Progressive Disease was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Event free estimates were determined using Kaplan-Meier estimates.
Time Frame: 6 Months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants | 17.0 [12.0 to 22.0] | 13.0 [8.0 to 18.0]

10. Secondary Outcome: Percentage of Participants With Disease Progression or Death in EGFR Positive and Negative Population (Data Cut Off 07 September 2010)
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR was determined by IHC.Tumor response was evaluated according to RECIST criteria (version 1.0). Progressive Disease was defined as At least a 20 % increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline, Weeks 3 and 6, Every 3 Weeks until Week 48 and Every 12 Weeks until Disease Progression or unacceptable toxicity up to 52 months
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 188 | 175
percentage of participants
  EGFR Positive (n=149,143) | 79.9 | 93.7
  EGFR Negative (n=39,32) | 89.7 | 90.6

11. Secondary Outcome: PFS in EGFR Positive and Negative Population (Data Cutoff 07 September 2010)
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR was determined by IHC. PFS was defined as time from randomization to the date of documented disease progression or death, whichever occurred first in EGFR positive and negative populations. Participants without progression were censored at the date of last tumor assessment where non progression was documented. If a participant receives a second anti-cancer therapy without prior documentation of disease progression, the participant was censored at the date of last tumor assessment before starting new chemotherapy. Kaplan-Meier estimates were used for analysis.
Time Frame: as for outcome 7
Population: FAS population; Only Participants with confirmed status of EGFR were included in the analysis; number of participants who were EGFR positive or negative
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 188 | 175
weeks
  EGFR Positive (n=149,143) | 8.9 [7.1 to 12.6] | 6.3 [6.1 to 7.3]
  EGFR Negative (n=39,32) | 11.5 [6.7 to 14.7] | 6.7 [5.9 to 12.0]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Comparison of EGFR positive populations; Test type: Superiority or Other; p = 0.0662, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.98 to 1.61]
Statistical Analysis 2: Comparison: Comparator vs Erlotinib; Comparison of EGFR negative populations; Test type: Superiority or Other; p = 0.9403, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.61 to 1.69]

12. Secondary Outcome: Probable Percentage of Participants Remaining Alive and Progression Free at 6 Months in EGFR Positive and Negative Population
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR was determined by IHC. Tumor response was evaluated according to RECIST criteria (version 1.0). PFS was defined as time from randomization to the date of documented disease progression or death, whichever occurred first in EGFR positive and negative populations. Participants without progression were censored at the date of last tumor assessment where non progression was documented. If a participant receives a second anti-cancer therapy without prior documentation of disease progression, the participant was censored at the date of last tumor assessment before starting new chemotherapy. Event free estimates were determined using Kaplan-Meier estimates.
Time Frame: 6 Months
Population: FAS population; n=number of EGFR positive or negative participants who remained at risk
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Comparator: Participants received either pemetrexed500 mg/m^2 every 21 days until disease progression, unacceptable toxicity or death or docetaxel 75 mg/m^2 every 3 weeks until disease progression, unacceptable t oxicity or death. Choice of comparator was left to the discretion of the investigator in countries where both treatments are registered to use and are commercially available for second line use (otherwise, docetaxel was administered), assigning the participant to either comparator depending upon the medical needs of the participant. Participants were required to receive concomitant treatment therapy as indicated in the product label.
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants
  EGFR Positive (n=23,18) | 20.0 [13.0 to 28.0] | 13.0 [7.0 to 19.0]
  EGFR Negative (n=4,5) | 11.0 [1.0 to 21.0] | 16.0 [3.0 to 29.0]

13. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of Confirmed Complete Response (CR) or Partial Response (PR) as Assessed by the Investigator Using RECIST
Description: Best overall response was defined as the best response according to RECIST recorded from the date of randomization until disease progression or recurrence. CR: disappearance of all target lesions; PR: reduction by at least 30% of the sum of the longest diameters of each target lesion, taking the initial sum of the longest diameters as a reference; Stable disease (SD): insufficient tumor reduction to define partial response and/or tumor increase less than that necessary to define tumor progression, taking as a reference the smallest sum of the longest diameter since the start of treatment; Progressive Disease (PD): increase by at least 20% in the sum of LD of each target lesion, taking as a reference the smallest sum of the longest diameters, reported since the start of treatment, or appearance of one or more new lesions. 95% Confidence Interval (CI) for one sample binomial using Pearson-Clopper method. Participants with a missing response were considered non-responders.
Time Frame: Baseline, Weeks 3 and 6, Every 3 Weeks until Week 48 and Every 12 Weeks until Disease Progression or unacceptable toxicity or Death or up to 52 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Erlotinib: Participants received a single oral dose of erlotinib 150 mg/day as a tablet until disease progression, unacceptable toxicity or death.
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 221 | 203
percentage of participants | 6.3 [3.5 to 10.4] | 7.9 [4.6 to 12.5]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.5349, Chi-squared — p-values are based on non-stratified analysis; Difference in Response Rates = 1.55, 95% CI 2-sided [-3.6 to 6.7] — Approximate 95% CI for the difference of two rates was determined using Hauck-Anderson Method

14. Secondary Outcome: Percentage of Participants With Deterioration in Quality of Life Determined Using Functional Assessment of Cancer Therapy - Lung (FACT-L)
Description: The FACT-L measures health related QOL and composes of five domains: the four domains (physical well being, emotional well being, social well being, functional well being) from the Functional Assessment of Cancer Treatment-General scale (FACT-G) and the lung cancer subscale (LCS). The FACT-L total score ranges from 0 to 136, higher scores represent better QOL.
Time Frame: as for outcome 10
Population: FAS population; Only participants with both a baseline FACT-L assessment and a subsequent FACT-L assessment were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 157
percentage of participants | 66.1 | 66.9

15. Secondary Outcome: Time to Deterioration in Quality of Life Using FACT-L
Description: The FACT-L measures health related QOL and composes of five domains: the four domains (physical well being, emotional well being, social well being, functional well being) from the FACT-G and the LCS. The FACT-L total score ranges from 0 to 136, higher scores represent better QOL. Time to deterioration of QoL or symptom progression is defined as time from randomization until either a clinically meaningful decline from baseline in Total FACT-L or, death on study, whichever occurs first. The clinically meaningful decline that was used to determine deterioration in QoL was ≥6-point decline from baseline. Participants without deterioration in QoL at the time of analysis were censored at the time of the last FACT-L assessment. Kaplan-Meier estimate was used to determine time to event.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 157
weeks | 9.0 [7.1 to 11.6] | 6.3 [6.1 to 8.0]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.1498, Log Rank; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.93 to 1.59]

16. Secondary Outcome: Probable Percentage of Participants Remaining Without Deterioration in Quality of Life at 6 Months as Assessed by FACT-L
Description: The FACT-L measures health related QOL and composes of five domains: the four domains (physical well being, emotional well being, social well being, functional well being) from the FACT-G and the LCS. The FACT-L total score ranges from 0 to 136, higher scores represent better QOL. Kaplan Meier estimates were used for analysis.
Time Frame: 6 Months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 157
percentage of participants | 25.0 [17.0 to 34.0] | 19.0 [11.0 to 26.0]

17. Secondary Outcome: Percentage of Participants With Symptomatic Progression Using FACT-L
Description: Participants' responses on the FACT-L were scored according to the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system manual. Time to symptom progression is the time from randomization until the earlier of a clinically meaningful decline from baseline in LCS score, or death on study. A change in 2 to 3 points on the LCS is a clinically meaningful change. Meaningful declines in scores as measured by the FACIT instruments have been found to be larger than improvements. Thus, deterioration in disease-related symptoms was defined by the upper bound (3 points) of the range of clinically meaningful change. However, participants who demonstrated early lung cancer progression demonstrated smaller changes from baseline score on the LCS. Therefore, the clinically meaningful decline that was used to determine progression of symptoms in this study was at least 1.5-point decline in LCS score from baseline.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
percentage of participants | 60.6 | 62.0

18. Secondary Outcome: Time to Symptomatic Progression Using FACT-L
Description: Participants' responses on the FACT-L were scored according to FACIT measurement system manual. Time to symptom progression is the time from randomization until the earlier of a clinically meaningful decline from baseline in LCS score, or death on study. A change in 2 to 3 points on the LCS is a clinically meaningful change. Meaningful declines in scores as measured by the FACIT instruments have been found to be larger than improvements. Thus, deterioration in disease-related symptoms was defined by the upper bound (3 points) of the range of clinically meaningful change. However, participants who demonstrated early lung cancer progression demonstrated smaller changes from baseline score on the LCS. Therefore, the clinically meaningful decline that was used to determine progression of symptoms in this study was at least 1.5-point decline in LCS score from baseline. Kaplan Meier estimated were used for analysis.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
weeks | 9.0 [7.0 to 12.1] | 7.1 [6.1 to 9.3]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.2202, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.90 to 1.57]

19. Secondary Outcome: Probable Percentage of Participants With Symptomatic Progression at 6 Months as Assessed by FACT-L
Description: as for outcome 18
Time Frame: 6 Months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
percentage of participants | 27 [18 to 36] | 27 [18 to 35]

20. Secondary Outcome: Percentage of Participants With Deterioration in the Trial Outcome Index (TOI)
Description: TOI is defined as the sum of the scores of the Physical Well- Being (PWB), Functional Well-Being (FWB), and LCS of the FACT-L instrument. Trial Outcome Index measures the physical functioning of participants. Time to deterioration in TOI is defined as time from randomization until the earlier of a clinically meaningful decline from baseline in TOI or death on study. The clinically meaningful decline used to determine deterioration in TOI was ≥6-point decline from baseline.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
percentage of participants | 60.0 | 63.3

21. Secondary Outcome: Time to Deterioration in the TOI
Description: TOI is defined as the sum of the scores of the PW, FWB, and LCS of the FACT-L instrument. Trial Outcome Index measures the physical functioning of participants. Time to deterioration in TOI is defined as time from randomization until the earlier of a clinically meaningful decline from baseline in TOI or death on study. The clinically meaningful decline used to determine deterioration in TOI was ≥6- point decline from baseline. Kaplan-Meier estimates were used for analysis.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
weeks | 9.3 [7.6 to 13.0] | 6.7 [6.1 to 9.4]
Statistical Analysis 1: Comparison: Comparator vs Erlotinib; Test type: Superiority or Other; p = 0.1063, Log Rank; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.95 to 1.66]

22. Secondary Outcome: Probable Percentage of Participants With Deterioration in the TOI at 6 Months as Assessed by FACT-L
Description: TOI is defined as the sum of the scores of the PW, FWB, and LCS of the FACT-L instrument. Trial Outcome Index measures the physical functioning of participants. Time to deterioration in TOI is defined as time from randomization until the earlier of a clinically meaningful decline from baseline in TOI or death on study. The clinically meaningful decline used to determine deterioration in TOI was ≥6-point decline from baseline. Kaplan-Meier estimates were used for analysis.
Time Frame: 6 Months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Comparator | Erlotinib
Number analyzed (Participants) | 165 | 158
percentage of participants | 28 [19 to 37] | 21 [13 to 29]

ADVERSE EVENTS:
Time Frame: All adverse events (related and unrelated) occurring during the study and for up to 28 days after the last dose of study medication were reported.
Description: All participants who received at least one dose of the trial medication and had at least one safety follow-up, whether withdrawn prematurely or not, were included in the safety analysis population (SAP).
Groups:
- Comparator: Participants received either Alimta 500 mg/m^2 every 21 days until disease progression, unacceptable toxicity or death or Taxotere 75 mg/m^2 every 3 weeks until disease progression, unacceptable toxicity or death. Choice of comparator was left to the discretion of the investigator in countries where both treatments are registered to use and are commercially available for second line use (otherwise, Taxotere was administered), assigning the participant to either comparator depending upon the medical needs of the participant. Participants were required to receive concomitant treatment therapy as indicated in the product label.
- Erlotinib: Participants received a single oral dose of erlotinib 150 mg/day until disease progression, unacceptable toxicity or death.
Arm/Group | Comparator | Erlotinib
Serious Adverse Events (participants affected / at risk) | 31/213 | 20/196
Other Adverse Events (participants affected / at risk) | 106/213 | 125/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator (N=213) | Erlotinib (N=196)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 0 | 1
Death (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator (N=213) | Erlotinib (N=196)
Rash (Skin and subcutaneous tissue disorders) | 7 | 74
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 12
Acne (Skin and subcutaneous tissue disorders) | 0 | 11
Diarrhoea (Gastrointestinal disorders) | 12 | 37
Nausea (Gastrointestinal disorders) | 29 | 15
Asthenia (General disorders) | 22 | 13
Fatigue (General disorders) | 18 | 9
Pyrexia (General disorders) | 14 | 10
Chest pain (General disorders) | 6 | 10
Oedema peripheral (General disorders) | 11 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Decreased appetite (Metabolism and nutrition disorders) | 22 | 17
Anaemia (Blood and lymphatic system disorders) | 16 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.